CLINICAL TRIAL: NCT06976567
Title: eUrologic Care in Nigeria: Increasing Access to Urologic Care for Rural Nigerians Using Telemedicine
Brief Title: Telemedicine for Urologic Care in Rural Nigeria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 25-43940
Record Dates: First submitted 2025-04-22; First posted 2025-05-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Urologic Disorders
Keywords: telemedicine; urologic care; health access
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group (Experimental): This group will engage in their urology consultation virtually.
  Interventions: Device: Telemedicine for urology consultations
- Standard of Care Group (No Intervention): This group will receive an in-person urologic consultation

INTERVENTIONS:
Device: Telemedicine for urology consultations — The patients that are assigned to the intervention group will receive a virtual urology consultation with urologists from Ahmadu Bello University in Zaria, Nigeria as opposed to physically presenting for the consultation.
  Other Names: Telemedicine Consultation
  Arms: Telemedicine Group

SUMMARY:
Access to urologic care in rural Nigeria is not as robust as it needs to be given the size of the population. This study will employ two research groups in rural Northern Nigeria. One group will receive urologic care via standard, in-person consultation. The second group will receive urologic care via telemedicine consultation. The main aim of this study is to assess whether telemedicine improves access to urologic care in these populations. Secondly, the investigators will assess patient satisfaction with their intervention via survey data.

DETAILED DESCRIPTION:
This is a multi-center study that will be using three primary care rural clinics in Kaduna State, Nigeria and a tertiary care hospital. These clinics were chosen based upon previous studies that have been conducted using them. Further, these sites were chosen for their relative frequency of patients presenting with urologic complaints. The clinics feature a primary doctor that fields urologic concerns and refers them to the main tertiary care center in Ahmadu Bello University in Zaria, Kaduna State, Nigeria. These clinics are in rural localities throughout the state, ensuring a broad representation of the study participant population.

Methods for telemedicine implementation have been discussed. The interventions will take place in the rural clinics and not at patients' homes given the clinics' reliable internet capabilities and for the consultations to be standardized. Our collaborators in Nigeria have been conducting an ongoing series of site visits to rural clinics in the proposed catchment area to assess for telemedicine capacity and any upgrades needed to make the rural clinics telemedicine capable.

The post-intervention survey will begin by collecting demographic variables such as age, gender, location of inhabitance, income, employment status, and ethnic group (due to the presence of many major and minor ethnic groups in Nigeria). Next, the survey will ask about patient experiences with ease of consultation, ease of travel, and the urologist's timeliness and responsiveness. Finally, the survey will ask about the cost and distance of travel for the urologic consultation, the time from initial presentation to the urology consultation, and patient satisfaction with care. A Likert scale will be employed for the ordinal variables, whereas patients will be able to manually enter estimates for continuous variables. Data from the RedCAP surveys will be securely stored in the research academic environment, allowing for data privacy.

Potential confounding variables, such as many of the demographic variables, will be addressed in the data analysis phase through stratification. Data will be analyzed using the appropriate statistical tests for the specific variables; Chi-squared or Fisher's exact tests will be used for categorical and binary variables, whereas T tests will be used for continuous variables. Multivariable generalized linear mixed effects regression models will be calculated with time to consultation as the primary outcome. The primary predictor in these models will be telemedicine consult compared to non-telemedicine consult. Potential confounding variables will be added including patient age, sex, location, ethnicity. Statistical significance will be defined by alpha > 0.05. All statistical testing will be completed using R and/or Stata.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old, any gender) that reside in rural Kaduna State.
* Present to primary clinics with an active urologic chief complaint(s), either surgical or non-surgical in nature.

Exclusion Criteria:

* Children (<18 years old).
* Individuals who do not live in rural Kaduna State localities.
* Those experiencing urologic emergencies.
* Those who do not present with any urologic chief complaints defined as the primary reason the patient is seeking medical care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time-to- Consultation | From enrollment to completion of post-consultation survey, which is 7 months.
  The time-to-urology consultation will be the primary outcome for this study. Essentially, the study will compare the time it takes for patients in either group to engage with a urologist. This measure was used in determining the power of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Bayne, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ahmadu Bello University, Zaria, Kaduna State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Muili AO, Mustapha MJ, Offor MC, Oladipo HJ. Emerging roles of telemedicine in dementia treatment and care. Dement Neuropsychol. 2023 May 29;17:e20220066. doi: 10.1590/1980-5764-DN-2022-0066. eCollection 2023. PMID 37261258
- [Background] Aronu NI, Atama CS, Chukwu NE, Ijeoma I. Socioeconomic Dynamics in Women's Access and Utilization of Health Technologies in Rural Nigeria. Community Health Equity Res Policy. 2022 Jan;42(2):225-232. doi: 10.1177/0272684X20972643. Epub 2020 Nov 26. PMID 33241987
- [Background] Doraiswamy S, Abraham A, Mamtani R, Cheema S. Use of Telehealth During the COVID-19 Pandemic: Scoping Review. J Med Internet Res. 2020 Dec 1;22(12):e24087. doi: 10.2196/24087. PMID 33147166
- [Background] Mahar JH, Rosencrance JG, Rasmussen PA. Telemedicine: Past, present, and future. Cleve Clin J Med. 2018 Dec;85(12):938-942. doi: 10.3949/ccjm.85a.17062. No abstract available. PMID 30526749
- [Background] Brimmo FO, Babatunde AO, Ezefuna NN, Kanu MS, Biziyaremye P. The need for more medical schools in medically underserved regions in Africa. Ann Med Surg (Lond). 2022 Nov 17;84:104967. doi: 10.1016/j.amsu.2022.104967. eCollection 2022 Dec. PMID 36426098
- [Background] Aslam MZ, Trail M, Cassell AK 3rd, Khan AB, Payne S. Establishing a sustainable healthcare environment in low- and middle-income countries. BJU Int. 2022 Feb;129(2):134-142. doi: 10.1111/bju.15659. Epub 2021 Dec 8. PMID 34837300
- [Background] Peters DH, Garg A, Bloom G, Walker DG, Brieger WR, Rahman MH. Poverty and access to health care in developing countries. Ann N Y Acad Sci. 2008;1136:161-71. doi: 10.1196/annals.1425.011. Epub 2007 Oct 22. PMID 17954679
- See also: Sample size calculation tool used to determine the study's sample size. — https://sample-size.net/sample-size-means/